CLINICAL TRIAL: NCT05484947
Title: The HIV Testing Trends and Outcomes at a Johannesburg Trauma ICU Unit
Status: Completed | Type: Observational
Sponsor: University of Witwatersrand, South Africa (Other)
Responsible Party: Principal Investigator, Maeyane Stephens Moeng, Professor, University of Witwatersrand, South Africa
Other Study IDs: Witwatersrand
Record Dates: First submitted 2022-07-23; First posted 2022-08-02 (Actual); Last update posted 2022-08-02 (Actual); Status verified 2022-07

CONDITIONS: Outcome, Fatal

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- HIV-positive: Those that were actually tested and had HIV-positive results
  Interventions: Diagnostic Test: Elisa HIV testing
- HIV-Negative: Those tested and had HIV-negative results
  Interventions: Diagnostic Test: Elisa HIV testing
- HIV-Unknown: those who had not volunteered for HIV testing

INTERVENTIONS:
Diagnostic Test: Elisa HIV testing — HIV testing on a voluntary basis
  Groups: HIV-Negative; HIV-positive

SUMMARY:
A retrospective observational study on the HIV testing trend and outcomes in a trauma population admitted to a critical care unit for care.

DETAILED DESCRIPTION:
Trauma ICU admission of 18 years and older were enrolled in the study. The HIV status was further divided into HIV-positive, HIV-negative, and HIV-unknown subgroups. The gender, ages, mechanism of injury, injuries sustained, ISS, physiological data, septic-related complications, and in-hospital mortality were noted and further analyzed.

Descriptive statistics were utilised using STATA version 15, and a p-value of <0.05 was considered statistically significant.

ELIGIBILITY:
Inclusion Criteria: Trauma patients admitted to a Trauma ICU at CMJAH -

Exclusion Criteria: Those under the age of 18 or with incomplete data

-

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Major Trauma patients admitted to a Trauma unit at a Johannesburg Trauma Unit
Sampling Method: Non-Probability Sample
Enrollment: 868 (Actual)
Dates: Start 2017-01-01 (Actual); Primary Completion 2018-12-31 (Actual); Study Completion 2021-08-18 (Actual)

PRIMARY OUTCOMES:
The HIV testing trends | study period over two years (from 01 January 2017 till 31 December 2018)
  Number tested for HIV in the study group
Outcomes | study period over two years (from 01 January 2017 till 31 December 2018)
  Septic related complications (wound infections, chest sepsis, septicaemia and sepsis related organ failure incidents

SECONDARY OUTCOMES:
Mortality | study period over two years (from 01 January 2017 till 31 December 2018)
  In-hospital mortality in the cohort

CONTACTS AND LOCATIONS:
Locations (1):
- Charlotte Maxeke Johanneburg Academic Hospital, Johannesburg, Gauteng, South Africa

IPD SHARING:
Plan to Share IPD: Undecided
only with close collaboration of future studies